CLINICAL TRIAL: NCT03001193
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Finding Study to Evaluate the Effect of Continuous Infusion of Tafoxiparin as an Adjunct Treatment to Oxytocin for up to 36 Hours in Term Pregnant, Nulliparous Women to Treat Primary Slow Progress of Labor Including Prolonged Latent Phase and Labor Arrest
Brief Title: Effect of Tafoxiparin to Treat Primary Slow Progress of Labor Including Prolonged Latent Phase and Labor Arrest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dilafor AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPL07
Record Dates: First submitted 2016-12-06; First posted 2016-12-22 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Labor, Obstetric
Keywords: Primary slow progress; Prolonged latent phase; Labor arrest
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DF01 low dose (Experimental): The subjects will receive intravenous infusion of DF01 (tafoxiparin) in low dose as an Adjunct Treatment to Oxytocin for up to 36 hours initiated by a pre-defined bolus dose as a therapeutic intervention until delivery
  Interventions: Drug: DF 01; Drug: Oxytocin
- DF01 medium dose (Experimental): The subjects will receive intravenous infusion of DF01 (tafoxiparin) in medium dose as an Adjunct Treatment to Oxytocin for up to 36 hours initiated by a pre-defined bolus dose as a therapeutic intervention until delivery
  Interventions: Drug: DF 01; Drug: Oxytocin
- DF01 high dose (Experimental): The subjects will receive intravenous infusion of DF01 (tafoxiparin) in high dose as an Adjunct Treatment to Oxytocin for up to 36 hours initiated by a pre-defined bolus dose as a therapeutic intervention until delivery
  Interventions: Drug: DF 01; Drug: Oxytocin
- PL1 (Placebo Comparator): The subjects will receive intravenous infusion of placebo as an Adjunct Treatment to Oxytocin for up to 36 hours initiated by a pre-defined bolus dose as a therapeutic intervention until delivery
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: DF 01
  Other Names: Tafoxiparin
  Arms: DF01 high dose; DF01 low dose; DF01 medium dose
Drug: Oxytocin
Drug: Placebo
  Other Names: PL1
  Arms: PL1

SUMMARY:
The study will be designed as a double-blind, placebo-controlled, parallel-group, dose-finding study with one group treated with placebo and three groups treated with tafoxiparin in three different infusion concentration levels, respectively. The intravenous infusion will be initiated by a pre-defined bolus dose infusion.

DETAILED DESCRIPTION:
Primary objective

To assess the dose-response relationship of tafoxiparin on the labor time defined as the time from the start of continuous infusion of tafoxiparin/placebo as an Adjunct Treatment to Oxytocin, until partus in term-pregnant, nulliparous women requiring labor augmentation due to Primary Slow Progress of Labor including prolonged latent phase and Labor Arrest.

Secondary objectives

To assess the safety and efficacy of tafoxiparin based on the safety and secondary efficacy parameters evaluated in the protocol. PK (pharmacokinetic) response in pregnant women during labor.

Methodology

All term-pregnant, nulliparous women presenting to the delivery ward are potential study patients unless they have already been enrolled in another clinical study. Subjects may be pre-informed about the study through the use of advertisements or information at the physician/midwife visits during pregnancy and at hospital admission.

The whole study includes the following steps:

* Screening and Baseline including informed consent and randomization
* Labor
* Discharge
* Follow-up at 8 (+/-1)weeks - End of study
* Safety follow up of infant at 6 months, +/-4 weeks, by telephone interview

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women of ≥18 to ≤45 years of age
2. Nulliparous
3. Gestational age > 36 weeks + 6 days confirmed by ultrasound
4. Experience slow progress of labor including prolonged latent phase and labor arrest (according to the respective definitions) etc

Exclusion Criteria:

1. Subjects with secondary slow progress or secondary labor arrest
2. BMI≥35 during first trimester of pregnancy
3. Breech presentation or other abnormal presentations etc

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 361 (Actual)
Dates: Start 2016-12; Primary Completion 2018-11 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Time from start of infusion of tafoxiparin/placebo until vaginal partus | Interval from start of study drug administration to vaginal delivery (hours, up to 36 hours )
  The primary endpoint (time from first infusion to vaginal partus) will be summarized graphically for each treatment group using Kaplan-Meier estimates. In addition to this statistical comparison between the treatments will be performed using the analysis of variance technique.

SECONDARY OUTCOMES:
Safety will be evaluated through rate and frequency of adverse events and serious adverse events | Through study completion ( 6 months, +/-4 weeks after delivery)
  Safety will be evaluated through rate and frequency of adverse events and serious adverse events, complete and symptom-directed physical evaluations, vital signs, safety blood samples (hematology and clinical chemistry), and rate of withdrawals from the study and/or the study medication
Time from cervical dilatation of 4 cm and progress of labor until vaginal partus | Interval from 4 cm of cervical dilatation to vaginal delivery (hours, up to 36 hours )
Proportion of women with dystocia/protracted labor defined as ≥8, 10, 12 and 14 hours of established labor (4 cm of cervical dilation to vaginal partus ) | Interval from 4 cm of cervical dilatation to vaginal delivery (hours, up to 36 hours )
Proportion of women with dystocia/protracted labor defined as ≥8, 10, 12 and 14 hours from start of study drug infusion to vaginal partus | Interval from start of study drug administration to vaginal delivery (hours, up to 36 hours )
Proportion of women with caesarean sections | From start of study drug administration to caesarean section (hours, up to 36 hours)
Proportion of women undergoing instrumental deliveries | From start of study drug administration to instrumental delivery (hours, up to 36 hours)
Use of analgesia (N2O, epidural, pudendal nerve block) | From start of study drug administration to any delivery (hours, up to 36 hours)
Proportion of women with postpartum hemorrhage > 1000 ml | From start of study drug administration and up to 7 days or discharge whichever comes first (days)
Fetal outcome measured as Apgar score (5 min) ≤ 7 points, Base Excess > -12 and referral to NICU (neonatal intensive care unit) (for > 48 hours | From start of study drug administration and up to 7 days or discharge whichever comes first (days)
Uterine hyperstimulation with fetal heart rate changes | From start of study drug administration to any delivery (hours, up to 36 hours)
Indication for referral to NICU | From start of study drug administration through study completion (6 months +- 4 weeks after delivery)
Use of Oxytocin (no. of mls. according to instructions) | From start of study drug administration to any delivery (hours, up to 36 hours)
Pharmacokinetic response | From start of study drug administration to any delivery (hours, up to 36 hours)
  Measurement of study drug in plasma at one time point

CONTACTS AND LOCATIONS:
Overall Officials: Gunvor Ekman-Ordeberg, MD, PhD, Study Chair — Dilafor AB
Locations (12):
- Hvidovre Hospital, Fødeafdelingen, Hvidovre, Denmark
- Finland (3):
  - Naistenklinikka (HUS) Naistentaudit ja synnytykset, Helsinki
  - Kätilöopiston Sairaala (HUS), Helsinki
  - Tampere University Hospital, Tampere
- Sweden (8):
  - Helsingborg Förlossningen, Helsingborgs Lasarett, Helsingborg
  - Länssjukhuset Ryhov, Jönköping
  - Karlstad Kvinnokliniken Centralsjukhuset, Karlstad
  - Kvinnokliniken Universitesjukhuset, Linköping
  - Kvinnokliniken Vrinnevisjukhuset, Norrköping
  - Skaraborgs sjukhus, Skövde
  - Norra Älvsborgs Länssjukhus, Trollhättan
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ekman-Ordeberg G, Hellgren-Wangdahl M, Jeppson A, Rahkonen L, Blomberg M, Pettersson K, Bejlum C, Engberg M, Ludvigsen M, Uotila J, Tihtonen K, Hallberg G, Jonsson M. Tafoxiparin, a novel drug candidate for cervical ripening and labor augmentation: results from 2 randomized, placebo-controlled studies. Am J Obstet Gynecol. 2024 Mar;230(3S):S759-S768. doi: 10.1016/j.ajog.2022.10.013. Epub 2023 May 17. PMID 38462256